CLINICAL TRIAL: NCT01791920
Title: Double-blinded, Randomized, Active Control Comparative, Multicenter-designed, Phase III Clinical Trial to Evaluate the Safety and Efficacy for Improvement of Glabellar Lines of "Botulax®" Compared to Botox Inj. in Patients With Moderate to Severe Glabellar Lines
Brief Title: To Evaluate the Safety and Efficacy of Botulax® Are Not Inferior to Those of Botox® in the Treatment of Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HG-11-01
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2013-02

CONDITIONS: Skin Aging
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin type A(Botox®) (Active Comparator): Botulinum toxin type A
  Interventions: Drug: Botulinum toxin type A(Botulax®)
- Botulinum toxin type A (Botulax®) (Experimental): Botulinum toxin type A
  Interventions: Drug: Botulinum toxin type A(Botox®)

INTERVENTIONS:
Drug: Botulinum toxin type A(Botulax®) — Single administration, Day 0, 20 units
  Arms: Botulinum toxin type A(Botox®)
Drug: Botulinum toxin type A(Botox®) — Single administration, Day 0, 20units
  Arms: Botulinum toxin type A (Botulax®)

SUMMARY:
To compare the safety and efficacy of Botulax® with Botox® in the improvement of moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 65
* Patients attaining grade 2 or 3 in the investigator's rating of glabellar lines severity at maximum frown
* Patients who voluntarily sign the informed consent
* Patients who can comply with the study procedures and visit schedule

Exclusion Criteria:

* Subjects who had facial plastic surgery (tissue augmentation, brow lift, and dermal resurfacing)treatment within 6 months. Those who had peeling or laser therapy
* Subjects with skin disorders, scar or infection around glabellar region
* Subjects who are taking Aspirin, NSAIDS or anti-coagulant
* Subjects with facial palsy or eyelid ptosis
* Subjects who diagnosed as neuromuscular junction disorder (e.g., myasthenia gravis, Lambert-Eaton Syndrome)
* Subjects with history of drug intoxication, alcohol abuse and/or depressive disorder
* Subjects with severe internal diseases (cardiovascular, respiratory, renal disease, liver disorder)
* Subjects who have previously been treated with botulinum toxin within 3 months (Botulinum toxin type A: 3months, type B: 4 months)
* Subject who have administered following drugs within the previous 4 months: Spectinomycin Hydrochloride, Aminoglycoside antibiotics, polypeptide antibiotics, tetracycline antibiotics, lincomycin antibiotics, muscle relaxants, anti-cholinergic agents, benzodiazepine and similar drugs, benzamide drugs, Tubocurarine-type muscle relaxants
* Subjects who have possibility to take the drugs listed above
* Subjects who have a plan to receive facial cosmetic procedures including dermal filler, chemical peeling and dermabrasion during study period
* Subjects who have glabellar lines that are unable to be improved with any physical method
* Subjects who have history of hypersensitivity to Botulinum toxin and other agents
* Subjects who are pregnant or breast-feeding
* Subjects who have a plan to be pregnant in 3months, or who are not doing contraceptive
* Subjects who participated in other studies within 30 days or were not passed over 5 times of half life for investigational product
* Subjects who are having trouble with acute disease
* Subjects who have taken any treatment that can affect to glabellar lines and/or any lines around forehead within the previous 6 months
* Subjects who are unable to communicate or follow the instructions
* Subjects who are not eligible for this study based on investigator's judgement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Responder rate of improvement in glabellar lines with Physician's rating of line severity | at 4 weeks post-injection
  Improvement rate of glabellar lines at maximum frown with Physician's rating of lines severity at 4weeks post injection.

SECONDARY OUTCOMES:
Safety evaluation in experimental drug treatment group | 4, 8, 12, 16 weeks post-injection
Responder rate of improvement in glabellar lines with Physician's rating of line severity | 8, 12, 16 weeks post-injection
  Improvement rate of glabellar lines at maximum frown with Physician's rating of lines severity at 8, 12, 16weeks post injection.
Responder rate of improvement in glabellar lines at rest with investigator's live assessment of severity | 4, 8, 12, 16 weeks post-injection
  Improvement rate of glabellar lines at rest with investigator's live assessment of severity at 4, 8, 12, 16weeks post injection
Responder rate of improvement in glabellar lines at maximum frown with investigator's photo assessment | 4, 8, 12, 16 weeks post-injection
  Improvement rate of glabellar lines at maximum frown with investigator's photo assessment at 4, 8, 12, 16weeks post injection
Responder rate of improvement in glabellar lines at rest with investigator's photo assessment | 4, 8, 12, 16 weeks post inejection
  Improvement rate of glabellar lines at rest with investigator's photo assessment at 4, 8, 12, 16weeks post injection
Responder rate of improvement in glabellar lines with Subject's improvement assessment | 4, 8, 12, 16 weeks post-injections
  Improvement rate of glabellar lines with Subject's improvement assessment at 4, 8, 12, 16weeks post injection
Subject's satisfaction rate | 4, 8, 12, 16 weeks post-injection
  Subject's satisfaction rate of improvement in glabellar lines at 4, 8, 12, 16 weeks post injection

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Chung-Ang University Hopspital, Seoul, Dongjak-gu
  - Seoul National University Hospital, Seoul, Jongno-Gu
  - National Medical Center, Seoul, Jung-Gu
  - Eulji General Hospital, Seoul, Nowon-Gu
  - The catholic university of Korea, Seoul ST. Mary's Hospital, Seoul, Seocho-Gu
  - Korea University Anam Hospital, Seoul, Seongbuk-Gu